CLINICAL TRIAL: NCT03304171
Title: Diet Quality Scores and Risk of Incident Breast Cancer in Healthy Women
Brief Title: Overall Diet Quality and Breast Cancer Risk
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Vikram Haridass, Principal Investigator, University of California, Irvine
Other Study IDs: 1998-453
Record Dates: First submitted 2017-10-03; First posted 2017-10-06 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Invasive Breast Cancer; Incident Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study was to examine the relationship between indices of overall diet quality and incident breast cancer risk in a large prospective cohort of women.

DETAILED DESCRIPTION:
This study examined the role of overall diet quality on the risk of developing invasive breast cancer among 96,959 women in the California Teachers Study, in which 4,826 women were diagnosed with breast cancer during follow-up (1995-2011). Participants' dietary habits were recorded at baseline (1995) using a 103-item Block95 Food Frequency Questionnaire to allow for the assessment of overall diet quality. Specifically, diet quality was characterized by the Alternate Mediterranean Diet (aMED), Alternative Healthy Eating Index-2010 (AHEI-2010), Dietary Approaches to Stop Hypertension (DASH), and Paleolithic Index scores. Associations between diet quality and the risk of developing breast cancer were examined using multivariate Cox proportional hazard regression models to provide hazard ratios and corresponding 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Participants with no history of cancer diagnosis prior to baseline.
* Participants with no history of myocardial infarction prior to baseline.
* Participants with no history of stroke prior to baseline.
* Participants with no history of diabetes prior to baseline.
* Participants who are not missing excessive dietary data.
* Participants with energy intake values at ≥1% and ≤99% of the population distribution.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Female participants of the California Teachers Study who met the eligibility criteria.
  The California Teachers Study is comprised entirely of female participants aged 22-104 years old at enrollment who were current and former public school teachers and administrators and completed a 16-page mailed questionnaire at study entry in 1995-1996. Details of the California Teachers Study (CTS) have been described previously (Bernstein L, et al.; 2002).
Sampling Method: Non-Probability Sample
Enrollment: 96959 (Actual)
Dates: Start 1995-10 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2011-12-31 (Actual)

PRIMARY OUTCOMES:
Incident Invasive Breast Cancer | 1995-2011
  All incident cancer cases were identified through linkage with the California Cancer Registry (CCR) records, which is a population-based cancer registry for California residents.

REFERENCES:
- [Background] Bernstein L, Allen M, Anton-Culver H, Deapen D, Horn-Ross PL, Peel D, Pinder R, Reynolds P, Sullivan-Halley J, West D, Wright W, Ziogas A, Ross RK. High breast cancer incidence rates among California teachers: results from the California Teachers Study (United States). Cancer Causes Control. 2002 Sep;13(7):625-35. doi: 10.1023/a:1019552126105. PMID 12296510
- See also: California Teacher Study Homepage — https://www.calteachersstudy.org/